CLINICAL TRIAL: NCT05660226
Title: Telemonitoring and E-Coaching in Hypertension
Acronym: TECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: Erasmus Medical Center (Other); Albert Schweitzer Hospital (Other); Sint Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 82758
Record Dates: First submitted 2022-11-08; First posted 2022-12-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
Keywords: Telemonitoring; Hypertension; E-Health; Coaching
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Home blood pressure monitoring + E-coaching
  Interventions: Other: Home blood pressure monitoring (telemonitoring)
- Control (Placebo Comparator): Standard care in patients with hypertension
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Home blood pressure monitoring (telemonitoring) — Using a digital mobile phone based telemonitoring platform to A: monitor patients and adjust their treatment accordingly based on the remote monitoring outcomes and B: provide E-Coaching/self learning modules (lifestyle)
  Arms: Intervention
Other: Standard care — Standard outpatient blood pressure management
  Arms: Control

SUMMARY:
Rationale: Hypertension is the most significant risk factor for cardiovascular disease and can be mitigated by lifestyle and medical management. Telemonitoring as a novel management approach to perform hypertension management at distance has been thriving but became indispensable during the COVID-19 pandemic. However, evidence of an effective implementation for telemonitoring remains to be elucidated.

Hypothesis: Telemonitoring with a smartphone application, which includes mixed automated services for a personal counselling program (PCP), on top of self-monitoring (SM) will lead to improvement of hypertension control rates, medication adherence and lifestyle behaviors and lower health care costs in patients with hypertension when compared to usual care.

Objective: To investigate the effects of PCP+SM on hypertension control rate and lifestyle behaviors as compared with usual care.

Study design: The study is a non-blinded randomized controlled clinical trial in adults with hypertension, in a multicenter hospital setting . We will randomize participants in a 1:1 fashion to the intervention group (PCP+SM), or to the control group (usual care).

Study population: 400 patients, patients, aged ≥18 years with hypertension (RR >140/90) Main study outcome: hypertension control rate (%<140/90mmHg) after 6 months (as measured by the SPRINT protocol)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hypertension (>140/90)
* Have and use a smartphone or a partner/caregiver who is able to provide the necessary technical support
* Able to provide written informed consent prior to participation in the study

Exclusion Criteria:

* Current user of a blood pressure monitor apporoved by the Dutch Heart foundation in combination with the Luscii app
* Persistent atrial fibrillation as indicated in the electronic health record (EHR)
* Pregnant or planning to become pregnant during the study period
* Severe kidney disease, defined as estimated glomerular filtration rate <30 per 1.73 m2 or currently on renal replacement therapy (i.e. hemodialysis or peritoneal dialysis)
* Unable to communicate (not language specific)
* Recent cardiovascular event (ischemic stroke, transient ischemic attack, myocardial infarction, coronary artery bypass grafting) in the past 3 months
* Diagnosis of dementia, psychosis as indicated in the electronic health record
* Life expectancy <1 year, for instance in terminal cancer or NYHA III or IV heart failure
* Individuals requiring BP monitor cuff size larger than 42cm
* Patients with proven secondary cause of hypertension for which drug treatment is not first choice (e.g. excessive licorice use, proven renal artery stenosis etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hypertension control rate | 6 months
  Percentage of patients with blood pressure on target (RR<135/85)

SECONDARY OUTCOMES:
Blood pressure control | 6 weeks, 6 months and 12 months
  Mean systolic and diastolic blood pressures for both groups
Medication use | 6 weeks, 6 months and 12 months
  Biochemical assessment of antihypertensive medication concentrations in blood. Number of antihypertensive agents used at 6 months. Number of antihypertensive medication changes at 6 months.
Self-management | baseline and 6 months
  Self-efficacy to monitor blood pressure, effect of coaching on disease insight and skills using PAM 13 and EQ5DL questionnaires
Patient and Healthcare provider Satisfaction | 6 months and 12 months
  Patients and health-care provider satisfaction as measured with TUQ and MAUQ questionnaires. The scales are from 1 to 7 (disagree to agree)
Hospitalizations | 6 months and 12 months
  Hospitalizations resulting from poor blood pressure control or cardiovascular complications resulting from poor blood pressure control (hypertensive emergencies, MI's, stroke)
Adverse cardiovascular events | 6 months and 12 months
  Myocardial infarction, cerebrovascular events and hypertensive emergencies.
Hypertension control rate | 6 weeks and 12 months
  Percentage of patients with blood pressure on target (RR<140/90)
Direct Medical Costs | 6 weeks, 6 months and 12 months
  * Costs related to HBPT (blood pressure monitor costs)
  * Costs related to additional prescribing of antihypertensive drugs
  * Costs related to a physical appointment for patients in a hypertension care pathway
  * Costs related to reimbursement for patients in a HBPT program
  * Costs related to hospital admissions resulting primarily from poorly controlled hypertension or hypertensive emergencies.
  * Costs related to hospital admissions or required care pathways following a cardiovascular complication as a result from poorly controlled hypertension
  * Future related medical costs
Direct Non-Medical Costs | 6 weeks, 6 months and 12 months
  * Training costs related to the use of HBPT for both telenurses, nurse specialists and clinicians
  * Development and exploitation costs (time spent developing the HBPT protocol, license costs for the application)
  * Salaries for involved health care providers during HBPT
Indirect Non-Medical costs | 6 weeks, 6 months and 12 months
  * Costs related to work absence (loss of productivity for short-term absence, friction cost for long-term absence)
  * Costs related to the hospital visit (travel costs, parking costs)
Indirect medical costs | 6 weeks, 6 months and 12 months
  o Future unrelated medical costs (as calculated using the iMTA PAID module: costs related to other diseases due to improved life expectancy

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Ziekenhuis, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No